CLINICAL TRIAL: NCT01495169
Title: A Multicenter, Open-label, Sequential Cohort, Dose-escalation, 14-day Study to Explore the Tolerability and Pharmacokinetics of Iloperidone 12 to 24 mg/Day Followed by 26 Weeks of Flexible Dosing (6 to 24 mg/Day) in Adolescent Patients (Aged 12 to 17 Years)
Brief Title: Tolerability and Pharmacokinetics of Iloperidone in Adolescent Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CILO522D2402
Record Dates: First submitted 2011-08-31; First posted 2011-12-19 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2016-06

CONDITIONS: Safety and Tolerability of Iloperidone
Keywords: Antipsychotic; Schizophrenia; Bipolar disorder; Iloperidone
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder | interventions — iloperidone; Tablets

ARMS (1):
- Iloperidone (Experimental): Part A (dose-escalation and fixed dose): Eligible patients receive iloperidone 2mg/day (1 mg BID) on day 1, then escalated every day for up to 12days utilizing a forced titration regimen to achieve a maximum dose of 12, 16, 20 or 24 mg/day given BID. Part B (optional extension phase): Patients who successfully complete Part A of the study are eligible to continue treatment with iloperidone for an additional 26 weeks
  Interventions: Drug: iloperidone (oral tablet)

INTERVENTIONS:
Drug: iloperidone (oral tablet) — iloperidone 12 to 24 mg/day followed by 26 weeks of flexible dosing (6 to 24 mg/day)

SUMMARY:
Tolerability, undertstanding of the action of the drug in the body, and understanding the effect of the drug in adolescent patients needing treatment with an antipsychotic medication

ELIGIBILITY:
Inclusion Criteria:

* males or females 12-17 years of age.
* in a stable housing situation with a guardian/parent who can encourage compliance with the study protocol.
* with diagnosis of disorder requiring treatment with an antipsychotic agent.
* having a Children's Global Assessment of Severity Scale (CGAS) of 41 or greater.
* Heart rate </=100 beats per minute and >/= 50 beats per minute.

Exclusion Criteria:

* Patients with mild, moderate or severe mental retardation (i.e., documented IQ <70), do not have the capacity to assent, cannot understand the informed consent, or participate fully in the assessments.
* Hospitalized due to suicidal ideation or suicidal behavior, history of suicidal ideation within 6 months prior to screening, history of suicidal behavior within 2 years prior to screening.
* Pregnant, females who can become pregnant and lactating females.
* Known hypersensitivity to iloperidone and to related drugs.
* Clinical conditions (Neurological, metabolic, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal or urological), which may pose significant risk to patients or impair reliable study participation.
* Clinically unstable cardiac disease, structural cardiac abnormalities, congential long QT syndrome, clinically significant ECG abnormalities at screening (PR interval >240 ms, QTcF >450 ms, QRS duration >/= 100 ms) or arrhythmias.
* Syncope, near syncope, or palpitations. Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2011-10; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of iloperidone at different dose levels based on AUC (area under the plasma concentration time curve during a dosage interval) Cmax ss (maximum plasma concentration at steady state), Tmax ss (time to Cmax at steady state). | Visit 5, 6, 7 (after at least 7 days of iloperidone treatment at the same dose level)
  Pharmacokinetics describes the action of a drug in the body over a period of time. Blood samples are collected to measure plasma concentrations of the study drug at different times after dosing. From the plasma concentration data, AUC, Cmax ss, and Tmax ss are calculated.
Tolerability of iloperidone at different dose levels | 14 days
  Frequency of treatment emergent adverse events, frequency of clinically notable changes from baseline in vital signs, electrocardiograms, laboratory tests, and reponses on movement disorder rating scales (Barnes Akathisia Rating Scale, Simpson-Angus Scale) and on a rating scale for suicidal thoughts and behaviors (Columbia Suicide Severity Rating Scale)

SECONDARY OUTCOMES:
Number of Patients with Adverse Events, Serious Adverse Events or Death | 26 weeks
  Safety and tolerability profile in open-label extension
Change from baseline in Clinical Global Impression of Improvement Scale (CGI-I) | Baseline, then Weekly for 2 weeks, then every 2-4 weeks for 26 weeks
  The CGI-I is scored from 1 to 7 and assesses the overall degree of illness relative to baseline. A CGI-I rating of 4 is equivalent to "no change." Ratings less than 4 are equivalent to "improvement" and ratings of more than 4 are equivalent to "worsening."
Change from baseline in the Children's Global Asessment Scale (CGAS | Baseline, then Weekly for 2 weeks, then every 2-4 weeks for 26 weeks
  The CGAS) is a numeric scale (1 through 100) used to rate the general functioning of children; high scores indicate better functioning.
Effect of iloperidone on QT, QT beat-to-beat (QTbtb), QT corrected using the Fridericia formulat (QTcF), QT corrected using the Bazett formula (QTcB), individual based correct QT (QTcI) | Baseline (24 hours), Visit 3 (4-hours post initial dose), and Visit 7 (13 hours
  Patients wear a holter monitor for ~24 hours during the baseline period, for an additional 4 hours after the first dose, and for ~13 hours after they have been on the same dose for at least 7 days to compare how the heart beats before and after the study drug is taken. The holter monitor transmits continuous data to a computer on how the heart beats for the time when the monitor is on and is a better measurement than data collected by a traditional electrocardiogram (ECG), which provides data on a limited number of heart beats over a short period of time.
Clinically notable changes from baseline on electrocardiogram (ECG) parameters (QTcF, QTcB, QRS, PR, heart rate) | Screening, baseline, 5x over 2 weeks, then every 2-4 weeks for 26 weeks
  Three ECGs are obtained for each assessment. The values are averaged for each ECG parameter (QTcF, QTcB, QRS, PR interval, heart rateare) and clinically notable changes from baseline and new or worsening heart rhythm disorders are identified

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (10):
- United States (10):
  - Novartis Investigative Site, Costa Mesa, California
  - Novartis Investigative Site, North Miami, Florida
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Coeur d'Alene, Idaho
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Marlton, New Jersey
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Cleveland, Ohio
  - Novartis Investigative Site, Salt Lake City, Utah